CLINICAL TRIAL: NCT07128082
Title: The Long COVID Treatment Trial
Acronym: LOCITT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Schmidt Initiative for Long COVID (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOCITT-T
Record Dates: First submitted 2025-08-14; First posted 2025-08-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 500 Participants will be randomized to receive placebo instead of active study medication. (Placebo Comparator)
  Interventions: Drug: Placebo
- 500 Participants will be randomized to receive active study medication. (Active Comparator)
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — The treatment group will receive the study medication (tirzepatide) for a 12 month period starting with a 2.5mg dose once a week.
  Arms: 500 Participants will be randomized to receive active study medication.
Drug: Placebo — Participants in the control group will receive a placebo instead of active study medication for a 12 month period.
  Arms: 500 Participants will be randomized to receive placebo instead of active study medication.

SUMMARY:
The goal of this study is to determine whether a medicine called tirzepatide, also called Zepbound, can reduce symptoms of Long COVID. A randomized control trial will allow us to measure the effect of the treatment by having half of the participants take the medication and half take a placebo that has no medication. Participants will take the medication (or placebo) they are given and complete study surveys for 12 months. All of the study tasks are done remotely from the comfort of a participants home.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older Living in the United States Able to read and understand English or Spanish Willing and able to participate in study interventions and activities, including;
* Access to an internet connected device
* Informed Consent
* Surveys
* Medication schedule
* Adverse Event reporting
* Weight reporting
* Use of wearable activity tracker
* Completing at home blood collections, if selected Meets the NASEM definition of Long COVID: an infection-associated chronic condition that occurs after SARS-CoV-2 infection and is present for at least 3 months as a continuous, relapsing and remitting, or progressive disease state that affects one or more organ systems 16.

Ability to verify identity Ability to verify diagnosis Agree to notify the study team if you start any other Long COVID treatments while enrolled in the study.

Complete the Fatigue Severity Scale with a minimum score of 36

Exclusion Criteria:

* Certain vulnerable populations (prisoners, children, fetuses, and institutionalized individuals)
* Women who are pregnant, excluded due to unknown risks to a fetus
* Personal or family history of medullary thyroid carcinoma
* History of severe gastrointestinal disease
* Diagnosis of gastroparesis
* Worsening or chronic renal failure
* History of pancreatitis
* Multiple Endocrine Neoplasia syndrome type 2
* Known serious hypersensitivity to tirzepatide
* Already taking tirzepatide or another GLP-1 agonist
* Medication contraindications to tirzepatide
* History of suicidal attempts and/or active suicidal ideation
* Underweight (BMI under 18.5)
* Planning to undergo elective surgery or procedures requiring general anesthesia or deep sedation in the next 12 months
* Symptoms of fatigue and/or brain fog that predated infection with COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Objective 1: Changes in fatigue severity score, measured by Fatigue Severity Scale (FSS) | 12 months
  The average difference in Fatigue Severity Scale (minimum score 9, maximum score 63, with higher scores indicating worse fatigue) between treatment and control groups of adults with Long COVID at month 3 or month 12 after study start

SECONDARY OUTCOMES:
Secondary Outcome: Changes in overall health, measured by European Quality of Life 5 day, 5 level (EQ-5D-5L) scores | 12 months
  EQ-5D-5L is a quality of life survey with a minimum score of 5 and a maximum score of 25, with a higher score indicating worse quality of life.
Secondary Outcome: Presence of and changes in post-exertional malaise, a condition that occurs in subsets of Long COVID and IACIs, measured by DePaul Symptom Questionnaire Post Exertional Malaise (DSQ-PEM) | 12 month
  DSQ-PEM evaluates the presence or absence of PEM and myalgic encephalomyelitis / chronic fatigue syndrome (ME/CFS)
Secondary Outcome: Changes in functional capacity as measured by Functional Capacity (FUNCAP) survey | 12 months
  The 27-question version of FUNCAP has a minimum score of 0 and a maximum score of 162, with a lower score indicating lower functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Moore Vogel, Principal Investigator — Scripps Translational Research Institute
Locations (1):
- Scripps Research, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
The investigators may share the coded study data with researchers outside of Scripps Research. Before doing so, they will ensure that nothing in the data can identify the participant directly.